CLINICAL TRIAL: NCT00434863
Title: A Comparative Randomized Double-Blinded Study of the Effect of Dysport and Botox on Forehead Wrinkles and EMG Activity
Brief Title: Comparative Study of the Effect of Dysport and Botox
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laserklinik Karlsruhe (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CR-015-LK/2005
Record Dates: First submitted 2007-02-12; First posted 2007-02-13 (Estimated); Last update posted 2007-02-13 (Estimated); Status verified 2007-02

CONDITIONS: Aging
Keywords: botulinum toxin type A; Dysport®; Botox®; hyperfunctional forehead lines; randomized controlled trial; double-blinded trial; electromyogram (EMG)
MeSH Terms: interventions — Botulinum Toxins, Type A

INTERVENTIONS:
Drug: botulinum toxin type A

SUMMARY:
The purpose of this study is to test the effect of Dysport and Botox on forehead wrinkles and EMG activity.

ELIGIBILITY:
Inclusion Criteria:

* age between 30 and 70 years
* moderate to severe hyperfunctional forehead wrinkles at maximum contraction and at rest

Exclusion Criteria:

* application of botulinum toxin products for a period of 12 months prior to the study
* any significant health disturbances
* facial nerve palsy, and any facial conditions that could confound safety or efficacy results
* pregnancy and breast-feeding
* neuromuscular diseases
* drugs interfering with neuromuscular function (e.g. aminoglycosides)

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2005-10; Study Completion 2006-03

PRIMARY OUTCOMES:
EMG Muscular Activity at baseline and 0.5, 1, 2, 4, 8 and 10 weeks after injection, followed by weekly examinations for a total observation period of 20 weeks
Frown Wrinkle Severity (photographs and questionnaire) at baseline and 0.5, 1, 2, 4, 8 and 10 weeks after injection, followed by weekly examinations for a total observation period of 20 weeks

SECONDARY OUTCOMES:
Side Effects upon completion of the study (20 weeks after injection)

CONTACTS AND LOCATIONS:
Overall Officials: Syrus Karsai, MD, Principal Investigator — Laserklinik Karlsruhe
Locations (1):
- Laserklinik Karlsruhe, Karlsruhe, Baden-Wurttemberg, Germany